CLINICAL TRIAL: NCT03214237
Title: A Cross-sectional Study of the Oral Health of Elderly Inpatients in Acute and Subacute Hospitals in Northumberland and North Tyneside
Status: Completed | Type: Observational
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ben J Steel, Dr Ben J Steel, Northumbria Healthcare NHS Foundation Trust
Other Study IDs: IRAS217606
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Oral Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Older adult inpatients on elderly care wards in acute hospitals within the Northumbria Hospitals NHS Foundation trust area, aged 70 or over and able to consent to involvement in the study
  Interventions: Other: no intervention - cross-sectional observational only

INTERVENTIONS:
Other: no intervention - cross-sectional observational only — no intervention - cross-sectional observational only

SUMMARY:
To provide a point-in-time measurement of the oral health of elderly inpatients across the trust (elderly defined here as over 70 years). This will provide information about the number of teeth, need for restorative and periodontal treatment, and extractions, the health of the oral mucosa, quality of any dentures and hygiene of the teeth and dentures.

DETAILED DESCRIPTION:
Such information will allow identification of any problems with oral health in this hospital population, thereby allowing development of strategies and protocols for managing these problems. There have been a number of studies examining these variables in elderly residents in care homes and a few in long term hospital settings (over 1 year admission), but only one in the UK previously in acute hospitals. Therefore the published literature is sparse, and requires further data collection. The oral health of the elderly, but particularly the institutionalized, is increasingly recognised for its important relationships with general health, wellbeing and quality of life. This study will provide useful information to address these concerns.

ELIGIBILITY:
Inclusion Criteria:

* age 70 or over and admitted to geriatric ward within the study area, able to consent

Exclusion Criteria:

* unable to consent, aged under 70

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: older adults admitted to elderly care wards within the trust. The hospital sites to be included are - NSECH, North Tyneside, Wansbeck, Hexham, Haltwhistle, Morpeth, Blyth, Alnwick and Berwick.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
level of oral hygiene | 1 month
  using modified plaque index

SECONDARY OUTCOMES:
age | 1 month
  age in years
gender | 1 month
  male or female
condition of oral mucosa | 1 month
  presence of absence of specific disease, e.g. candidosis, leukoplakia
number of broken and decayed teeth | 1 month
  a simple count of the number of decayed and broken teeth present

CONTACTS AND LOCATIONS:
Overall Officials: Ben J Steel, Principal Investigator — Northumbria Hospitals NHS Foundation Trust
Locations (1):
- Northumbria Hospitals NHS, Cramlington, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not planned to be shared